CLINICAL TRIAL: NCT02504177
Title: Clinical Trial for Optimal Novel Oral Anticoagulant (NOAC) Schedule Immediate Before Catheter Ablation for Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0387
Record Dates: First submitted 2015-07-14; First posted 2015-07-21 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The group of keep medication NOAC (Experimental): The randomization after scheduling of Ablation at clinic The explanation to stop taking medicine of NOAC 24 hours before the ablation
  Interventions: Drug: novel oral anticoagulant for 30 days
- The group of stop medication NOAC 1 day (Active Comparator): The randomization after scheduling of ablation at clinic. The explanation to stop taking medicine of NOAC day of ablation
  Interventions: Drug: novel oral anticoagulant for 24 hour

INTERVENTIONS:
Drug: novel oral anticoagulant for 30 days — novel oral anticoagulant includes 'dabigatran,Pradaxa®', 'rivaroxaban,Xarelto®', and 'apixaban, Eliquis®'.
  Arms: The group of keep medication NOAC
Drug: novel oral anticoagulant for 24 hour — novel oral anticoagulant includes 'dabigatran,Pradaxa®', 'rivaroxaban,Xarelto®', and 'apixaban, Eliquis®'.
  Arms: The group of stop medication NOAC 1 day

SUMMARY:
This study is to evaluated the interruption schedule of NOAC in patients who undergo atrial fibrillation ablation. The investigators will compare the bleeding complications were classified as major and minor bleeding, thromboembolic, vascular complications, Re-admission and increased in the length of hospital stay during the 30-day post-radiofrequency catheter ablation(RFCA) period among patients who interrupt NOAc 24hours before ablation and patients who stop NOAC in the morning of the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who consent with study
2. Patients with Atrial fibrillation (20-80 years old)
3. patients who undergoing catheter ablation of atrial fibrillation due to symptomatic, drug refractory atrial fibrillation
4. Patients possible to NOAC

Exclusion Criteria:

1. Patients who do not agree with study inclusion
2. eGRF < 30ml/min
3. Impossible to NOAC
4. Structural cardiac disease
5. Major hemorrhagic complication
6. CHA2DS2-VASc score > 5
7. Patients who have experienced Ischemic cerebellar infarction more than 2times

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
incidence of major bleeding complications | during 30 days post-AF ablation.
  Bleeding complication is assessed by physical examination or laboratory measurement

SECONDARY OUTCOMES:
incidence of thromboembolism | during 30 days post-AF ablation.
  thromboembolism is diagnosed by both clinical situations and image studies combined.
incidence of minor bleeding | during 30 days post-AF ablation.
Re-admission rate related procedure | during 30 days post-AF ablation.
length of hospital stay | during 30 days post-AF ablation.
incidence of vascular complications | during 30 days post-AF ablation.
  vascular complication is diagnosed by both clinical situations and image studies combined.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea